CLINICAL TRIAL: NCT06884995
Title: Correlation of Weight Loss With Residual Gastric Volume and Shape on Computerized Tomography in Patients Undergoing Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mahmoud alazawy, lecteurer of general surgery, Helwan University
Other Study IDs: helwan university 84-2024
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Weight Regain Post Bariatric Surgery
Keywords: shape, Sleeve gastrectomy, inadequate weight loss, volumetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 20 patients had sleeve gastrectomy: after 12 months ,volumetry study was done

SUMMARY:
Laparoscopic sleeve gastrectomy (LSG) has been accepted as a primary bariatric procedure. The aim of the study was to evaluate the volume and the morphologies of remnant stomachs after LSG and their association with weight loss

DETAILED DESCRIPTION:
Twenty patients who underwent Laparoscopic sleeve gastrectomy (LSG) were followed prospectively and evaluated at 12 months after operation using computed tomography CT with 3D reconstruction to evaluate the shape and volume of the residual stomach after LSG. Total sleeve volume (TSV), tube volume (TV), antral volume (AV) and tube/antral volume ratio (TAVR) were included.

ELIGIBILITY:
Inclusion Criteria:

* candidate for sleeve gastrectomy

Exclusion Criteria:

* revisional surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Twenty patients who underwent Laparoscopic sleeve gastrectomy (LSG) were followed prospectively and evaluated at 12 months after operation using computed tomography CT with 3D reconstruction to evaluate the shape and volume of the residual stomach after LSG
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-07-07 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
volume of sleeve and shape | 12 months
  relation with weight loss

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided